CLINICAL TRIAL: NCT05420311
Title: Personalized or Precision Medicine in the Dietary Approach to Obesity
Acronym: PI21/01677
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PI21/01677
Record Dates: First submitted 2022-05-18; First posted 2022-06-15 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-04

CONDITIONS: Obesity
Keywords: Precision medicine, nutrigenomics, microbiome, obesity, diet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: A randomized cross-over study testing three different dietary weight-loss interventions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A balanced hypocaloric diet in macronutrients (MedDiet). (Experimental): Mediterranean diet based on olive oil as main fat and regular consumption of vegetables (2 daily rations), fruits (3 daily rations), legumes (3 weekly rations), fish (3 weekly rations), with low consumption of red meat and meat products (less than twice a week), dairy foods (less than once a week) and no sweets, pastries or sugary drinks. Diet will produce a 600 kcal per day caloric deficit, according to the Harris-Benedict equation for each subject. Diet will include 45% carbohydrates, 35% fat, 20% protein distributed in at least 4 meals (breakfast, lunch, afternoon snack and dinner).
  Interventions: Other: MedDiet Arm
- A very low carbohydrate diet (KetoDiet). (Experimental): Diet will produce a 600 kcal per day caloric deficit, according to the Harris-Benedict equation for each subject. Diet will include 5 % carbohydrates, 65% fat and 30% high biological value protein
  Interventions: Other: KetoDiet Arm
- An intermittent fasting (IF) approach. (Experimental): In this diet subjects alternate norm caloric diet during 24 h (according to Harris-Benedict equation) and a diet including only 25% of caloric requirements the following 24 h (this day diet will include 5 % carbohydrates, 65% fat and 30% high biological value protein).
  Interventions: Other: IF Arm

INTERVENTIONS:
Other: MedDiet Arm — A balanced hypocaloric diet in macronutrients (MedDiet)
  Arms: A balanced hypocaloric diet in macronutrients (MedDiet).
Other: KetoDiet Arm — A very low carbohydrate diet (KetoDiet).
  Arms: A very low carbohydrate diet (KetoDiet).
Other: IF Arm — An intermittent fasting (IF) approach
  Arms: An intermittent fasting (IF) approach.

SUMMARY:
The main objective of this project is to apply a precision medicine approach to try to explain the intra-individual variability of the response to different weight loss approaches: a balanced hypocaloric diet in macronutrients (MedDiet), a very low carbohydrate diet (KetoDiet) and an intermittent fasting (IF) approach, and try to establish in a personalized manner with the individual variability in genetics, metabolites, intestinal microbiome, and environmental factors the best dietary strategy for weight loss. As secondary objectives the investigators pretend to O1: To analyze whether individual variability in genetics, epigenetics, intestinal microbiome, and environmental factors determine the changes in insulin resistance, blood pressure, lipid levels and NASH markers after three different dietary interventions. O2: To analyze whether individual variability in genetics, epigenetics, intestinal microbiome, and environmental factors determine the changes in the body composition and the different ratio of free-fat/ fat mass loss after three different dietary interventions. O3: To determine the most effective intervention to increase the loss of fat mass, preserve the free-fat mass and trigger a better metabolic profile. O4: To follow-up changes in gut microbiota and DNA methylation after each of the cross-over dietary interventions. O5: To evaluate the transcriptional response of adipose tissue and elucidate its predictive value for the body-composition changes in patients subjected to the different dietary interventions.

O6: To evaluate the influence of D-ß-hydroxybutyrate as well as other short-chain acyl-CoA precursor metabolites in human adipocytes lipolysis by in vitro experimentation and elucidate the influence of metabolite-sensitive histone modifications in the shaping of adipose transcriptional program and lipolysis sensitivity. O7: To develop a machine learning algorithm based on genetics, epigenetics, intestinal microbiome, and environmental factors for the prediction of the best dietary approach for weight loss in a personalized manner. To try to respond to these objectives, the investigators will apply two models: a randomized cross-over study testing three different dietary weight-loss interventions: MedDiet, KetoDiet, and IF with wash-out periods before each intervention.

DETAILED DESCRIPTION:
The main objective of this project is to apply a precision medicine approach to try to explain the intra-individual variability of the response to different weight loss approaches: a balanced hypocaloric diet in macronutrients (MedDiet), a very low carbohydrate diet (KetoDiet) and an intermittent fasting (IF) approach, and try to establish in a personalized manner with the individual variability in genetics, metabolites, intestinal microbiome, and environmental factors the best dietary strategy for weight loss. As secondary objectives the investigators pretend to O1: To analyze whether individual variability in genetics, epigenetics, intestinal microbiome, and environmental factors determine the changes in insulin resistance, blood pressure, lipid levels and NASH markers after three different dietary interventions. O2: To analyze whether individual variability in genetics, epigenetics, intestinal microbiome, and environmental factors determine the changes in the body composition and the different ratio of free-fat/ fat mass loss after three different dietary interventions. O3: To determine the most effective intervention to increase the loss of fat mass, preserve the free-fat mass and trigger a better metabolic profile. O4: To follow-up changes in gut microbiota and DNA methylation after each of the cross-over dietary interventions. O5: To evaluate the transcriptional response of adipose tissue and elucidate its predictive value for the body-composition changes in patients subjected to the different dietary interventions. O6: To evaluate the influence of D-ß-hydroxybutyrate as well as other short-chain acyl-CoA precursor metabolites in human adipocytes lipolysis by in vitro experimentation and elucidate the influence of metabolite-sensitive histone modifications in the shaping of adipose transcriptional program and lipolysis sensitivity. O7: To develop a machine learning algorithm based on genetics, epigenetics, intestinal microbiome, and environmental factors for the prediction of the best dietary approach for weight loss in a personalized manner. To try to respond to these objectives, the investigators will apply two models: a randomized cross-over study testing three different dietary weight-loss interventions: MedDiet, KetoDiet, and IF with wash-out periods before each intervention in patients with obesity; and a second cellular approach with adipose tissue from the patients as well as with commercial cells.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 18 and <70 years old who were derived to the obesity-management unit of the Endocrinology and Nutrition Unit of the Virgen de la Victoria Hospital (Málaga).
* BMI between 35 and 45 kg/m2.

Exclusion Criteria:

* Pregnant or lactating
* Following a prescribed diet for any reason in the past 3 months
* Celiac disease, Crohn's disease or any condition altering nutritional requirements.
* Allergies or food intolerances, as well as antibiotics treatment or usual probiotics intake.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-10-31 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight after each intervention | From baseline to 1 month
  Weight in kg

SECONDARY OUTCOMES:
Changes in body composition and in the ratio of free-fat / fat mass loss after the three different dietary interventions. | From baseline to 1 month
  Ratio in %
Changes in the degree of insulin resistance. | From baseline to 1 month
  Measured by the HOMA-IR ratio
Changes in the systolic blood pressure | From baseline to 1 month
  Blood pressure measured in millimeters of mercury
Changes in the diastolic blood pressure | From baseline to 1 month
  Blood pressure measured in millimeters of mercury
Changes in lipid profile (triglycerides) | From baseline to 1 month
  Measured in mg/dl
Changes in lipid profile (cholesterol) | From baseline to 1 month
  Measured in mg/dl
Changes in the degree of ketosis | From baseline to 1 month
  Measured in mmol/l
Changes in gut microbiota | From baseline to 1 month
  Change from baseline in 16S rRNA amplicons after 1 month
DNA methylation. | From baseline to 1 month
  Measured by a Methylation Array of the whole genome interrogating 850000 CpGs.
Changes in the punctuation in neurocognitive test - Trailmaking Test (A - B) | From baseline to 1 month
  Trailmaking Test (A - B) allows evaluating visual search speed, working memory, motor skills, visual-spatial sequencing, sustained attention, divided attention and mental flexibility (time: reduction in seconds)
Changes in the punctuation in neurocognitive test - Stroop | From baseline to 1 month
  Stroop measures selective attention and inhibitory control. (increasing scores)
Changes in the punctuation in neurocognitive test - WAISspan | From baseline to 1 month
  Letters and numbers from the WAISspan for working memory, concentration, auditory sequencing and executive attention. (time: reduction in seconds)
Changes in the punctuation in neurocognitive test - UPPS-P | From baseline to 1 month
  * Trailmaking Test (A - B) allows evaluating visual search speed, working memory, motor skills, visual-spatial sequencing, sustained attention, divided attention and mental flexibility (time: reduction in seconds)
  * Stroop: Measures selective attention and inhibitory control. (increasing scores)
  * Letters and numbers from the WAISspan for working memory, concentration, auditory sequencing and executive attention. (time: reduction in seconds)
  * UPPS-P: Impulse BehaviorScale (Cyders et al. 2007; validated in Spanish by Candido et al, 2012). Self- administered scale that evaluates impulsivity. Scale of items using a 4-point likert scale (min 59 /max 136 points).

CONTACTS AND LOCATIONS:
Overall Officials: Franscisco J. Tinahones, MD, PhD., Principal Investigator — Instituto de Investigacion Biomedica de Malaga
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain